CLINICAL TRIAL: NCT00265551
Title: A Randomized, Double-Blind, Placebo-Controlled, Olanzapine-Referenced, Parallel Group Safety, Efficacy, and Tolerability Study of SCA-136 in Subjects With Acute Exacerbations of Schizophrenia
Brief Title: Study Evaluating SCA-136 in Subjects With Acute Exacerbations of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3153A1-202
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

INTERVENTIONS:
Drug: SCA-136 (200 mg)
Drug: SCA-136 (400 mg)
Drug: olanzapine (15 mg)
Drug: placebo

SUMMARY:
The purpose of this study is to determine whether a low dose and a high dose of the study drug SCA-136 are effective and safe in the treatment of schizophrenia requiring hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia
* Ability to remain hospitalized for at least first 4 weeks of study
* Needs hospitalization due to worsening of schizophrenia

Exclusion Criteria:

* Type 1 or 2 diabetes
* Previous use of clozapine
* Serious medical illness other than schizophrenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2006-01; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to day 42 on the positive subscale of the SCI-PANNS

SECONDARY OUTCOMES:
Change from baseline to day 42 on:
SCI-PANNS total score
negative symptom sub-scale score of SCI-PANNS
general psychopathology subscale score of SCI-PANNS
response rate based upon SCI-PANNS total score
BPRS score
CGI-S score
CGI-I score
Cognitive assessments scores

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (32):
- United States (32):
  - Little Rock, Arkansas
  - Cerritos, California
  - Costa Mesa, California
  - La Mesa, California
  - Oceanside, California
  - Paramount, California
  - Pico Rivera, California
  - Rosemead, California
  - San Diego, California
  - Torrance, California
  - Middletown, Connecticut
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Kissimmee, Florida
  - North Miami, Florida
  - Hoffman Estates, Illinois
  - Indianapolis, Indiana
  - Lake Charles, Louisiana
  - Baltimore, Maryland
  - Rockville, Maryland
  - St Louis, Missouri
  - Willingboro, New Jersey
  - Cedarhurst, New York
  - Holliswood, New York
  - Chagrin Falls, Ohio
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Fort Washington, Pennsylvania
  - Memphis, Tennessee
  - Austin, Texas
  - DeSoto, Texas
  - Tacoma, Washington

REFERENCES:
- [Derived] Shen JH, Zhao Y, Rosenzweig-Lipson S, Popp D, Williams JB, Giller E, Detke MJ, Kane JM. A 6-week randomized, double-blind, placebo-controlled, comparator referenced trial of vabicaserin in acute schizophrenia. J Psychiatr Res. 2014 Jun;53:14-22. doi: 10.1016/j.jpsychires.2014.02.012. Epub 2014 Feb 24. PMID 24613032